CLINICAL TRIAL: NCT04501393
Title: Recommended Clear Fluid Intake Volume at 2 Hours Prior to Esophagogastroduodenoscopy for Adult Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 382/2563
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 ml/kg (No Intervention): The participants will not be asked to drink anything at 2 hours prior to planned procedure.
- 3 ml/kg (Active Comparator): The participants will be asked to drink 3ml/kg of clear liquid at 2 hours prior to planned procedure.
  Interventions: Other: Clear liquid intake
- 7 ml/kg (Active Comparator): The participants will be asked to drink 7 ml/kg of clear liquid at 2 hours prior to planned procedure.
  Interventions: Other: Clear liquid intake
- 10 ml/kg (Active Comparator): The participants will be asked to drink 10 ml/kg of clear liquid at 2 hours prior to planned procedure.
  Interventions: Other: Clear liquid intake

INTERVENTIONS:
Other: Clear liquid intake — Clear oral fluid including water, pulp-free juice and tea or coffee without milk
  Arms: 10 ml/kg; 3 ml/kg; 7 ml/kg

SUMMARY:
Research in developing patient fasting guidelines was developed years ago. On a physiological basis, patients with a longer fasting time may have less residual gastric content and lower risk of pulmonary aspiration. The recent Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration of The American Society of Anesthesiologists (ASA) was published in March 2017. Current practice consists of 2-hour fasting period for clear oral fluid (including water, pulp-free juice and tea or coffee without milk), 4- hour fasting period for breast milk and 6-hour fasting period for non-human milk and solid food. However, there are only few supportive and suggestive scientific evidences. The purpose of this study is to evaluate the current clinical practice guidelines for preoperative fasting to enhance the quality of pediatric anesthesia care and promote patient safety.The investigators plan to enroll adults aged 18-60 years, who are scheduled for esophago-gastro-duodenoscopy (EGD), in order to study the effects of fasting time and the actual intragastric volume which may help us establish a comprehensive fasting guideline.

DETAILED DESCRIPTION:
Research in developing patient NPO guidelines was developed years ago. On a physiological basis, patients with a longer fasting time may have less residual gastric content and lower risk of pulmonary aspiration. The recent Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration of The American Society of Anesthesiologists (ASA) was published in March 2017. Current practice consists of 2-hour fasting period for clear oral fluid (including water, pulp-free juice and tea or coffee without milk), 4- hour fasting period for breast milk and 6-hour fasting period for non-human milk and solid food. However, there are only few supportive (category A) and suggestive (category B) scientific evidences.

Since Maltby et al showed results of patient's safety in elective surgical patients who had clear oral fluid intake 2 hours before surgery in 1986, the published clinical evidence is still insufficient to address the relationship between pulmonary aspiration and fasting time . For breast milk, infant formula and solid food, the latest Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration in 2011 also follow previous suggestion of fasting time because of inadequate updated supportive clinical trials.

The purpose of this study is to evaluate the current clinical practice guidelines for preoperative fasting to enhance the quality of pediatric anesthesia care and promote patient safety. Andersson et al. reviewed 10,015 pediatric anesthesia charts retrospectively and found an incidence of 3 cases of pulmonary aspiration in 10,000 pediatric anesthesia patients who were allowed to drink clear liquid fluids until called to operative rooms . This approach promotes patient safety by minimizing a patient's dehydration status and reduced intraoperative hypotensive events. Furthermore, shortened fasting times also decreases patient irritability and improves parental satisfaction in preoperative experiences.

The investigators plan to enroll adults ages 18-60 years old, who are scheduled for esophago-gastro-duodenoscopy (EGD) at Siriraj hospital. This observational study will be conducted in 2 stages; (1) preoperative period (2) intraoperative period. Patients' demographic information will be collected along with NPO history including times, volume and type of fluid/ food intake in the preoperative period. Intragastric volume and pH from each patient's stomach at the beginning of EGD procedure will be measured in the intraoperative period.

The investigators believe that the information from this study will help us understand the effects of NPO time and the actual intragastric volume which may help establish a comprehensive NPO guideline.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18-60 years scheduled for EGD procedure
* Patient who willing to participate in this study

Exclusion Criteria:

* Patient who scheduled for emergent EGD procedures
* Patients with active upper GI bleeding
* Patients who received preoperative oral medication
* BMI > 30 kg/m2
* Patients with previous GI motility or acid-base pathology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Residual gastric volume | at 2 hour after drinking, during endoscopic procedure
  Collect actual intra-gastric content volume after drinking assigned amount of fluid at 2-hour fasting period of each patient.

SECONDARY OUTCOMES:
Gastric acidity (pH) | at 2 hour after drinking, during endoscopic procedure
  Collect actual intra-gastric content pH after drinking assigned amount of fluid at 2-hour fasting period of each patient.
Hypotension | at 2 hour after drinking, during endoscopic procedure
  Compare hypotension incidence of each group
Post operative nausea and vomitting | pre-endoscopic procedure
  Compare postoperative nausea and vomiting incidence of each group
Ready to discharge time | When the procedure finish until ready to discharge, approximately 1-2 hours after endoscopy
  Compare ready to discharge time of each group

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No